CLINICAL TRIAL: NCT01821859
Title: A Phase II Evaluation of Abraxane Plus Bevacizumab for the Treatment of Recurrent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Abraxane/Bevacizumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low enrollment
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00005859
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Ovarian Cancer; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Albumin-Bound Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abraxane/Bevacizumab (Experimental): Bevacizumab will be infused at a dose of 10 mg/kg in 100 mL normal saline over 30 minutes ± 10 minutes. It is given first, prior to the Abraxane infusion.
  Abraxane will be infused at a dose of 220 mg/m² in 20 mL normal saline per 100 mg vial over 30 minutes. This will follow the Bevacizumab infusion.
  Interventions: Drug: Abraxane; Drug: Bevacizumab

INTERVENTIONS:
Drug: Abraxane — Abraxane will be infused at a dose of 220 mg/m² in 20 mL normal saline per 100 mg vial over 30 minutes. This will follow the Bevacizumab infusion.
Drug: Bevacizumab — Bevacizumab will be infused at a dose of 10 mg/kg in 100 mL normal saline over 30 minutes ± 10 minutes. It is given first, prior to the Abraxane infusion.

SUMMARY:
The protocol will study the effect of the combination of two drugs-Abraxane and Bevacizumab-on a subject's ovarian cancer, fallopian tube cancer, or primary peritoneal cancer. This study drug combination will be given to subjects who have already been treated for their cancer with other chemotherapy, and now their cancer has become worse or has come back again. Neither one of these study drugs has been approved by the FDA for treatment in these three types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma. Histologic documentation of the original primary tumor is required via the pathology report.
* All patients must have measurable disease. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be >20mm when measured by conventional techniques including CT, and MRI, or >10 mm when measured by spiral CT.
* Patients must have at least one "target lesion" to be used to assess response as defined by RECIST. Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy.
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment.
* Patients are required to receive at least one additional cytotoxic regimen for management of recurrent or persistent disease. Patients are allowed to receive, but are not required to receive, biologic (non-cytotoxic) therapy either alone or as part of the cytotoxic regimens for management of recurrent or persistent disease.
* Age >18 years. Women all races and ethnic groups will be included.
* Patients with an ECOG performance status < 2. ( see APPENDIX A)
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count >1,500/uL
* platelets >100,000/uL
* hemoglobin >9 g/dL
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
* Alkaline Phosphatase within normal institutional limits
* creatinine <1.5 X institutional upper limit of normal
* Neurologic function: Neuropathy (sensory and motor) less than or equal to CTCAE v4.0 grade 2. (see APPENDIX B)
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 28 days prior to entering the study or whose adverse events due to agents administered more than 28 days earlier continue to be grade 3 or greater.
* Patients may not have received any other investigational agents within the past 28 days.
* Any hormonal therapy or immunotherapy directed at the malignant tumor must be discontinued at least one week prior to enrollment. Continuation of hormone replacement therapy is permitted. Continuation of other established medical treatments for a known medical condition is permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Abraxane or Bevacizumab.
* Patients who have had prior therapy with Abraxane.
* Patients who have received radiation to more than 25% of marrow-bearing areas. (see APPENDIX C)
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last five years.
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last five years are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than five years prior to registration, and the patient remains free of recurrent or metastatic disease.
* Patients who have known active liver disease or hepatitis.
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
* Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
* Patients with clinically significant cardiovascular disease, including:

uncontrolled hypertension, myocardial infarction, unstable angina within 6 months of enrollment, NYHA Grade II or greater heart failure, serious cardiac arrhythmia requiring medication, grade II or greater peripheral vascular disease.

* Patients with clinically significant proteinuria. Patients with a urine protein of 1+ on dipstick should undergo a 24-hour urine collection, which must demonstrate < 100 mg protein/24 hr to allow participation in the study.
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
* Patients who have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment on the study, or anticipation of need for major surgical procedure during the course of the study.
* Patients who have received commercial bevacizumab within 28 days prior to enrollment on the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection(with the exception of uncomplicated UTI), chronic non- healing wound, bone fracture, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded from this study because of possible risk to the fetus or infant.
* Known HIV-positive patients are excluded from the study because of possible risk of lethal infection when treated with marrow suppressive therapy.
* Safety data regarding Abraxane use in patients with ascites is not available; therefore patients with symptomatic ascites will be excluded from participation in the study. Patients may have asymptomatic ascites.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Pejovic, MD, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Abraxane/Bevacizumab: Bevacizumab will be infused at a dose of 10 mg/kg in 100 mL normal saline over 30 minutes ± 10 minutes. It is given first, prior to the Abraxane infusion.
  Abraxane will be infused at a dose of 220 mg/m² in 20 mL normal saline per 100 mg vial over 30 minutes. This will follow the Bevacizumab infusion.
  Bevacizumab : Bevacizumab will be infused at a dose of 10 mg/kg in 100 mL normal saline over 30 minutes ± 10 minutes. It is given first, prior to the Abraxane infusion.
  Abraxane : Abraxane will be infused at a dose of 220 mg/m² in 20 mL normal saline per 100 mg vial over 30 minutes. This will follow the Bevacizumab infusion.
Period: Overall Study
Arm/Group | Abraxane/Bevacizumab
Started | 5
Completed | 0
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Abraxane/Bevacizumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival Rate at 6 Months as Defined as Complete Response, Partial Response, or Stable Disease.
Description: Using RECIST criteria, Complete Response (CR)= disappearance of all target lesions, Partial Response (PR)= At least a 30% decrease in the sum of the longest diameter of target lesions, and Stable Disease (SD)= neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as progressive disease.
Time Frame: 6 months after start of dosing
Arm/Group | Abraxane/Bevacizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Abraxane/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes